CLINICAL TRIAL: NCT02785380
Title: Laparoscopic Surgery Versus Radiofrequency Ablation for the Treatment of Recurrent Hepatocellular Carcinoma
Brief Title: Laparoscopic Surgery VS RFA for Recurrent HCC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Military Medical University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Ph.D.,M.D., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC007
Record Dates: First submitted 2016-05-25; First posted 2016-05-27 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic surgery(LS) (Experimental): For LS,the patient was usually placed in the lithotomy position. Pneumoperitoneum was maintained at a pressure between 12 and 14 mmHg.Intra-operative ultrasonography was performed routinely. Large bile duct branches or vessels were clipped before division and minor hemostasis was carried out using bipolar diathermy. Large hepatic vein branches were divided by endovascular staplers. The Pringle maneuver was not used. Wedge resection, segmentectomy or subsegmentectomy was performed. The surgeon aimed to achieve a 1.0-cm safety margin during the liver resection.
  Interventions: Procedure: laparoscopic surgery(LS)
- Radiofrequency ablation(RFA) (Active Comparator): RFA was performed according to the Guidelines of Radiofrequency Ablation Therapy for Liver Cancer: Chinese Expert Consensus Statement issued by the Chinese Society of Liver Cancer and Chinese Society of Clinical Oncology. RFA was performed by using a commercially available Cool-tipTM RFA system (Valleylab, Boulder, CO, USA), or a RF 2000 system (Radio-Therapeutics Mountain View, CA).
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: laparoscopic surgery(LS) — For LS, the patient was usually placed in the lithotomy position. Pneumoperitoneum was maintained at a pressure between 12 and 14 mmHg. Three to 4 working ports sized between 5 mm and 12 mm were used . Intra-operative ultrasonography was performed routinely. Parenchymal transection was performed using a Cavitron ultrasonic surgical aspirator (CUSA, Valleylab, Boulder, CO, USA). Large bile duct branches or vessels were clipped before division and minor hemostasis was carried out using bipolar diathermy. Large hepatic vein branches were divided by endovascular staplers. A 1.0-cm safety margin was planed to get during the liver resection.
  Arms: laparoscopic surgery(LS)
Procedure: RFA — RFA was performed according to the Guidelines of Radiofrequency Ablation Therapy for Liver Cancer: Chinese Expert Consensus Statement issued by the Chinese Society of Liver Cancer and Chinese Society of Clinical Oncology RFA was performed under real-time ultrasound guidance. RFA was performed by using a commercially available Cool-tipTM RFA system (Valleylab, Boulder, CO, USA), or a RF 2000 system (Radio-Therapeutics Mountain View, CA). Grounding was achieved by attaching 2 pads to the patient's back or legs.
  Arms: Radiofrequency ablation(RFA)

SUMMARY:
Management of recurrent HCC is urgent and several treatments have been developed .Repeat hepatectomy is considered to be the first choice for recurrent HCC.

Unfortunately, repeated open hepatectomy can be performed only in a small proportion of patients due to inadequate liver function reserve, widespread recurrence or high invasiveness. Given that recurrent tumors are usually detected at small size during follow-up after initial surgery, radiofreqency ablation (RFA), which is less invasive, may be locally curative and causes minimal damage to liver function reserve,has been widely used. However, the re-recurrence rate after RFA is more than 50%,and the recurrence-free survival is less than 20%. Recently, satisfactory short- and long-term oncological outcomes have been reported for laparoscopic surgery (LS) for the treatment for primary HCC with cirrhosis. Some single center pilot studies reported that LS may, compared with open surgery, improve the prognosis of HCC with less blood loss and shorter hospital stay. LS was initially considered not suitable for recurrent HCC due to postoperative adhesions that might make laparoscopic surgical procedure more difficult and less safe. With improvement in technique and experience, recent studies showed that LS for recurrent HCC in cirrhotic patients is a safe and feasible procedure with good short-term outcomes. However, thus far, no study has been performed to evaluate the long-term oncological outcomes of LS for recurrent HCC, and compare those results to that for RFA. To clarify these issues, a multicenter retrospective comparative study by using propensity score matching method that included a large consecutive series of patients with recurrent HCC within Milan criteria, who underwent LS or RFA, was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. First recurrent HCC after curative hepatectomy;
3. A solitary recurrent HCC ≤ 3.0 cm in diameter, or multiple recurrent HCC ≤ 3 lesions, each ≤ 3.0 cm in diameter;
4. Tumor located in left lateral lobe (segment II or III) or subcapsule of liver(subcapsular nodule was defined as a lesion located less than 1 cm from the liver edge and could be treated by either LS or RFA.
5. No radiologic evidence of invasion into major portal/ hepatic vein branches;
6. No extrahepatic metastases;
7. Child-Turcotte-Pugh class A or B;

Exclusion Criteria:

1. Coagulation disorders (prothrombin activity <40% or a platelet count of <80,000/mm3);
2. History of hepatic encephalopathy, ascites refractory to diuretics or esophageal or gastric variceal bleeding;
3. History of a secondary malignancy;
4. Severe dysfunction of the heart, kidney, or other organs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years

OTHER OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Background] Camma C, Di Marco V, Orlando A, Sandonato L, Casaril A, Parisi P, Alizzi S, Sciarrino E, Virdone R, Pardo S, Di Bona D, Licata A, Latteri F, Cabibbo G, Montalto G, Latteri MA, Nicoli N, Craxi A; Unita Interdipartimentale Neoplasie Epatiche (U.I.N.E) Group. Treatment of hepatocellular carcinoma in compensated cirrhosis with radio-frequency thermal ablation (RFTA): a prospective study. J Hepatol. 2005 Apr;42(4):535-40. doi: 10.1016/j.jhep.2004.11.042. PMID 15868653
- [Background] Poon RT, Fan ST, Lo CM, Liu CL, Wong J. Intrahepatic recurrence after curative resection of hepatocellular carcinoma: long-term results of treatment and prognostic factors. Ann Surg. 1999 Feb;229(2):216-22. doi: 10.1097/00000658-199902000-00009. PMID 10024103